CLINICAL TRIAL: NCT01646164
Title: Effect of Dill Seed on Uterus Contractions Pattern
Status: Completed | Type: Observational
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Samira Ebrahimzadeh Zagami, MUMS, Mashhad University of Medical Sciences
Other Study IDs: Effect of Dill seed
Record Dates: First submitted 2012-07-18; First posted 2012-07-20 (Estimated); Last update posted 2012-07-20 (Estimated); Status verified 2012-07

CONDITIONS: Uterus Contractions Pattern
Keywords: Dill seed; Pattern of uterus contractions; Active phase of labor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Dill seed: used dill seed infusion (1 tablespoon whole dill seed seeped in a half or whole cup boiling water for 3-4 min)
- No used Dill seed: those who had not used any herbal drugs were placed at the control group

SUMMARY:
Dill is herbaceous and aromatic herb used in order to convenient and shorter labor in Iran. The objective of this study was to evaluate the effect of Dill seed on uterus contractions in active phase of labor.

ELIGIBILITY:
Inclusion Criteria:

* 18-35 yrs, primiparous, having single fetus with cephalic presentation, gestational age 37-42 weeks, having no medical diseases, having no history of hospitalization due to psychological diseases, having no addiction to cigarette, having no complications during pregnancy such as hypertension, and BMI< 26.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: pregnance women
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2009-05; Primary Completion 2010-06 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Dill seed | up to 15 months
  used dill seed infusion (1 tablespoon whole dill seed seeped in a half or whole cup boiling water for 3-4 min)